CLINICAL TRIAL: NCT06321315
Title: The Effect of Case-based Teaching on Critical Thinking Motivation, Motivation and Knowledge Acquisition in Midwifery Undergraduate Students
Brief Title: The Effect of Case-based Teaching on Midwifery Undergraduate Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Esra KARATAŞ OKYAY, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KSUESRAKARATASOKYAY006
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Midwifery Students
Keywords: Case discussion; Motivation; Critical thinking; Obtaining information; Midwifery; Student

STUDY DESIGN:
Intervention Model Description: Intervention group (Case-based instruction group) Control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Case-based instruction group) (Experimental): Case-based teaching will be provided to second-year students who take the risky pregnancy and care course for the first time, who are included in the case-based teaching group by randomization method.
  Interventions: Behavioral: Case-based instruction
- Control (No Intervention): The control group is the group in which no intervention was made.

INTERVENTIONS:
Behavioral: Case-based instruction — Case-based instruction will be applied to the students in the intervention group. "Student Information Form", "Critical Thinking Motivation Scale", "Academic Motivation Scale" and "Knowledge Assessment Form" will be . All students will receive classical in-class theoretical education about such as hemorrhages, hyperemesis gravidarum, oligohydramnios and urinary system diseases. In the intervention group, after the theoretical teaching of each subject within the scope of the Risky Pregnancy and Care course, cases prepared on the basis of the subject taught to the students will be applied. "Student Information Form (13th and 14th questions)", "Critical Thinking Motivation Scale", "Academic Motivation Scale", "Knowledge Assessment Form" and "Visual Comparison Scale" will be applied to all students as post-test data after case-based teaching of four topics.
  Arms: Intervention group (Case-based instruction group)

SUMMARY:
Case-based teaching will be applied to second year midwifery undergraduate students. The intervention group (case-based teaching implementation group) and the control group each consist of 35 students.

DETAILED DESCRIPTION:
Materials and Methods: The randomized controlled study will be conducted between March-April 2024 with 70 students (35 intervention group and 35 control group) who are studying in the second year of Kahramanmaraş Sütçü İmam University, Faculty of Health Sciences, Department of Midwifery and taking the risky pregnancy and care course for the first time. Case-based teaching will be applied to the students in the intervention group. The students will be informed about the method to be followed in the study, the voluntary information form will be read to those who want to participate in the study, and their verbal and written permissions will be obtained. "Student Information Form", "Critical Thinking Motivation Scale", "Academic Motivation Scale" and "Knowledge Assessment Form" will be applied to the students as pre-test data with face-to-face method before the classical theoretical education in the classroom. Classical in-class theoretical education will be given to all students on the most frequently encountered risky pregnancy diagnoses such as hemorrhages, hyperemesis gravidarum, oligohydramnios and urinary system diseases. In the intervention group, the cases prepared on the basis of the subject taught to the students after each subject will be applied after the theoretical teaching of each subject within the scope of the Risky Pregnancy and Care course. The application will take place on different days, in 4 sessions and in each session, case-based teaching will be done for different topics. Each application is expected to last approximately 60-100 minutes. The cases in question were created by the researchers by reviewing the literature. The students in the control group will not be given any application after the classical theoretical education in the classroom. "Student Information Form (13th and 14th questions)", "Critical Thinking Motivation Scale", "Academic Motivation Scale", "Knowledge Assessment Form" and "Visual Comparison Scale" will be applied to all students as post-test data after the case-based instruction of four subjects.

ELIGIBILITY:
Inclusion Criteria:

* Who agreed to participate in the research,
* 2nd year midwifery student taking the "Risky Pregnancy and Care" course,
* No clinical experience in hemorrhages, hyperemesis gravidarum, oligohydramnios and urinary system diseases (Health Vocational High School Graduate etc.).

Exclusion Criteria:

* Incomplete completion of data collection forms,
* Not participating in all case-based teaching phases,
* Who want to leave the study,
* Working as a midwife in any health institution,
* Who have taken this course before.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Determination of Critical Thinking Motivation | At the first interview, the Critical Thinking Motivation Scale was applied to all students in both groups as a pre-test
  The Critical Thinking Motivation Scale (CTMS) consists of 19 items and is rated on a Likert-type scale from 1 to 6. It has two main sub-dimensions as "expectancy" and "value". Consisting of 4 items, the main sub-dimension "expectation" aims to measure individuals' perceptions of the possibility of accomplishing the tasks. The second main sub-dimension, "value", has 15 items. The main sub-dimension "Value" consists of "achievement" (4 items), "usefulness" (4 items), "intrinsic value/interest value" (4 items) and "compensation" (3 items) The first sub-dimension of the main sub-dimension "Value", "achievement", measures the importance of doing a task well; "intrinsic value" measures the pleasure derived from doing a task; "usefulness" refers to how a task fits with one's future plans; "cost" refers to the constraint that engaging in an activity places on other activities, the evaluation of how much effort is required to complete the activity, and the emotional cost of doing so.
Determination of Critical Thinking Motivation | Four weeks after the first interview, the Critical Thinking Motivation Scale is administered as a pre-test to all students in both groups.
  The Critical Thinking Motivation Scale (CTMS) consists of 19 items and is rated on a Likert-type scale from 1 to 6. It has two main sub-dimensions as "expectancy" and "value". Consisting of 4 items, the main sub-dimension "expectation" aims to measure individuals' perceptions of the possibility of accomplishing the tasks. The second main sub-dimension, "value", has 15 items. The main sub-dimension "Value" consists of "achievement" (4 items), "usefulness" (4 items), "intrinsic value/interest value" (4 items) and "compensation" (3 items) The first sub-dimension of the main sub-dimension "Value", "achievement", measures the importance of doing a task well; "intrinsic value" measures the pleasure derived from doing a task; "usefulness" refers to how a task fits with one's future plans; "cost" refers to the constraint that engaging in an activity places on other activities, the evaluation of how much effort is required to complete the activity, and the emotional cost of doing so.

SECONDARY OUTCOMES:
Determining the level of Academic Motivation | At the first interview, the Academic motivation scale was applied to all students in both groups as a pre-test
  The academic motivation scale was developed by Bozanoğlu in 2004. Consisting of 20 items, the scale is 5-point Likert type. Students mark the items according to their suitability (1= Absolutely not suitable, 5= Absolutely suitable). The score range in the scale is 20-100. The higher the score on the scale, the higher the academic motivation of the individual.
Determining the level of Academic Motivation | Four weeks after the first interview, the Academic motivation scale is administered as a pre-test to all students in both groups.
  The academic motivation scale was developed by Bozanoğlu in 2004. Consisting of 20 items, the scale is 5-point Likert type. Students mark the items according to their suitability (1= Absolutely not suitable, 5= Absolutely suitable). The score range in the scale is 20-100. The higher the score on the scale, the higher the academic motivation of the individual.
Determining the status of access to information | At the first interview, the information assessment form was applied to all students in both groups as a pre-test
  It is a multiple-choice questionnaire form created by the researchers after an extensive literature review in order to evaluate the knowledge of the students taking the Risky Pregnancy and Care course about the topics taught in case-based teaching. This question form was created in line with the learning objectives of the "Risky Pregnancy and Care" course. The draft form was revised after the expert opinion evaluation of the case examples and appropriate corrections and additions were made. After the revision of the case examples, the draft form of the revised information assessment form was submitted to the experts in the field of midwifery for evaluation in terms of comprehensibility, inclusiveness, expression and language. After the necessary revision, it will be applied as a multiple-choice pre- and post-test. The highest score of the form is 100 and the lowest score is 0 (max=100, min=0).
Determining the status of access to information | Four weeks after the first interview, the information assessment form is administered as a pre-test to all students in both groups.
  It is a multiple-choice questionnaire form created by the researchers after an extensive literature review in order to evaluate the knowledge of the students taking the Risky Pregnancy and Care course about the topics taught in case-based teaching. This question form was created in line with the learning objectives of the "Risky Pregnancy and Care" course. The draft form was revised after the expert opinion evaluation of the case examples and appropriate corrections and additions were made. After the revision of the case examples, the draft form of the revised information assessment form was submitted to the experts in the field of midwifery for evaluation in terms of comprehensibility, inclusiveness, expression and language. After the necessary revision, it will be applied as a multiple-choice pre- and post-test. The highest score of the form is 100 and the lowest score is 0 (max=100, min=0).
Evaluation of satisfaction with the training methods used and the effect of training methods on perceptions of competence during clinical practice | At the first interview, the Visual Comparison Scale was applied to all students in both groups as a pre-test
  It was used to assess students' satisfaction with the training methods used and the effect of the training methods on their perception of competence during clinical practice. In the scale, 0 means "not at all satisfied" and 10 means "very satisfied".
Evaluation of satisfaction with the training methods used and the effect of training methods on perceptions of competence during clinical practice | Four weeks after the first interview, the Visual Comparison Scale is administered as a pre-test to all students in both groups.
  It was used to assess students' satisfaction with the training methods used and the effect of the training methods on their perception of competence during clinical practice. In the scale, 0 means "not at all satisfied" and 10 means "very satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Esra KARATAŞ OKYAY, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
we don't share individual participant data with other researchers

REFERENCES:
- [Background] Gholami M, Changaee F, Karami K, Shahsavaripour Z, Veiskaramian A, Birjandi M. Effects of multiepisode case-based learning (CBL) on problem-solving ability and learning motivation of nursing students in an emergency care course. J Prof Nurs. 2021 May-Jun;37(3):612-619. doi: 10.1016/j.profnurs.2021.02.010. Epub 2021 Mar 2. PMID 34016321
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34016321/